CLINICAL TRIAL: NCT02924428
Title: Clinical Evaluation of Venus Versa Diamonpolar Applicator Treatment Followed by AC Dual Applicator Treatment Using 2 Intense Pulsed Light Wavelength Bands for Facial Acne Vulgaris
Brief Title: Venus Versa Diamondpolar Applicator Treatment Followed by AC Dual Applicator Treatment for Facial Acne Vulgaris
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not commenced
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS2715
Record Dates: First submitted 2016-09-30; First posted 2016-10-05 (Estimated); Results first posted 2020-10-14 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-10

CONDITIONS: Acne Vulgaris
Keywords: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diamondpolar applicator, AC Dual applicator (Experimental): Radio frequency (RF) and pulsed magnetic field (PEMF) treatment followed by intense pulsed light (IPL) treatment delivered to the skin using the Venus Versa system.
  The RF and PEMF applicator has 4 electrodes which emit RF and PEMF simultaneously.
  The IPL applicator operates a blue light (415 nm) and also red light (630 nm) simultaneously. The IPL applicator also includes a sapphire cooled light guide of 10x30mm.
  Interventions: Device: Venus Versa
- AC Dual applicator treatment (Active Comparator): Intense pulsed light (IPL) treatment delivered to the skin using the Venus Versa system.
  The IPL applicator operates a blue light (415 nm) and also red light (630 nm) simultaneously. The IPL applicator also includes a sapphire cooled light guide of 10x30mm.
  Interventions: Device: Venus Versa

INTERVENTIONS:
Device: Venus Versa

SUMMARY:
The purpose of the study is to evaluate the efficacy of facial acne vulgaris treatment using the Venus Versa Diamondpolar applicator in combination with the Venus Versa AC dual applicator using two intense pulsed light wavelength bands.

DETAILED DESCRIPTION:
Multi-center, prospective, open-label study utilizing before-after study design. Up to 20 healthy subjects, age 18 - 55 years with acne vulgaris who wish to improve their skin appearance will be randomized to receive either Diamondpolar applicator (radio frequency and pulsed magnetic field) treatment followed by AC Dual applicator (intense pulsed light) treatment or AC Dual applicator (intense pulsed light) treatment alone using the Venus Versa system. Duration of subject participation will be approximately 10 weeks (4 weekly treatments with a follow-up visit scheduled 6 weeks after the last treatment).

The AC Dual applicator (IPL) is indicated for the treatment of acne vulgaris by using a blue light (415 nm) to target porphyrins produced by the P. acne bacteria, destroying the bacteria and uses the red light (630 nm) to help reduce inflammation, inhibit sebum production and improve healing.

The addition of the Diamondpolar applicator (RF and PEMF) treatment is thought to target the sebaceous gland, causing it to shrink and decrease sebum output

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick skin phototype I - VI
* Having mild to moderate acne vulgaris (as defined by the Acne Global Severity Scale) and have at least 10 inflammatory and 15 non-inflammatory lesions, but no nodulo-cystic lesions.
* Subject who can commit to all treatments and follow up.

Exclusion Criteria:

* Superficial metal or other implants in the treatment area.
* Current or history of cancer, or current condition of any type of cancer, or pre-malignant moles.
* Pregnancy and nursing.
* Patients with cystic acne, acne conglobata, acne fulminans, or secondary acne (chloracne, drug-induced acne, etc)
* Diseases which may be stimulated by light at the wavelengths used, such as history of Systemic Lupus Erythematosus, Porphyria, and Epilepsy.
* Patients with history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treatment area, may be treated only following a prophylactic regimen.
* Poorly controlled endocrine disorders, such as Diabetes or Polycystic Ovary Syndrome.
* Any active condition in the treatment area, such as sores, Psoriasis, eczema, and rash.
* Tattoos, scars or piercings in the treated area.
* History of skin disorders, keloids, abnormal wound healing, as well as very dry and fragile skin.

  • Use of medications, herbs, food supplements, and vitamins known to induce photosensitivity to light exposure at the wavelengths used, such as Isotretinoin (Accutane) within the last six months, tetracyclines, or St. John's Wort within the last two weeks.
* Any surgical procedure in the treatment area within the last three months or before complete healing.
* Treating over tattoo or permanent makeup.
* Excessively tanned skin from sun, tanning beds or tanning creams within the last two weeks.
* As per the practitioner's discretion, refrain from treating any condition which might make it unsafe for the patient.
* Exposure to investigational product within 3 months (or designated half-life) prior to enrollment.
* Prior drugs, interventions, skin laser/light or another device for Acne treatment within 3 months of initial treatment or during the course of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2016-09; Primary Completion 2018-06-05 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph L Reiz, Study Director — Venus Concept Ltd.
Locations (1):
- Sadick Research Group, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eight patients signed the consent form but did not meet inclusion/exclusion criteria.
Groups:
- AC Dual Applicator: Intense pulsed light (IPL) treatment delivered to the skin using the Venus Versa system.
  The IPL applicator operates a blue light (415 nm) and also red light (630 nm) simultaneously. The IPL applicator also includes a sapphire cooled light guide of 10x30mm.
Period: Overall Study
Arm/Group | Diamondpolar Applicator, AC Dual Applicator | AC Dual Applicator
Started | 20 | 19
Completed | 16 | 14
Not Completed | 4 | 5
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 2 | 4
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diamondpolar Applicator, AC Dual Applicator | AC Dual Applicator | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 19 | 39
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 33
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 17 | 14 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 14 | 13 | 27
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Baseline Inflammatory and Non-inflammatory Lesions [Mean (Standard Deviation); unit: Lesions] — Average baseline count of number of inflammatory and non-inflammatory acne lesions per treatment group.
  Lesions
    Inflammatory Lesions | 7.25 (5.30) | 6.95 (4.24) | 7.10 (4.78)
    Non-inflammatory Lesions | 13.9 (8.18) | 11.05 (6.96) | 12.51 (7.69)

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Acne Vulgaris Appearance
Description: Treatment will be considered successful if the appearance improves by at least 2 points on the 5-point Global Acne Assessment Score (GAAS) at 6 weeks post treatment as compared to baseline where 0 = No evidence of facial acne vulgaris, 1 (minimal) = Few non-inflammatory lesions (comedones) are present; a few inflammatory lesions (papules/pustules) may be present, 2 (mild) = Several to many non-inflammatory lesions (comedones) are present; a few inflammatory lesions (papules/pustules) are present, 3 (Moderate) = Many non-inflammatory (comedones) and inflammatory lesions (papules/pustules) are present; no nodulo-cystic lesions are allowed, 4 (Severe) = Significant degree of inflammatory disease; papules/pustules are a predominant feature; a few nodulo-cystic lesions may be present; comedones may be present. Lower number represents an improvement in acne vulgaris.
Time Frame: Week 10 (6 weeks after last treatment)
Population: This primary outcome measurement will not be evaluated as data was not collected.
Arm/Group | Diamondpolar Applicator, AC Dual Applicator | AC Dual Applicator
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Reduction of Inflammatory Lesions and Non-inflammatory Lesions
Description: Reduction in the number of inflammatory lesions and non-inflammatory lesions counted on treatment area
Time Frame: Week 10 (6 weeks after last treatment)
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Diamondpolar Applicator, AC Dual Applicator | AC Dual Applicator
Number analyzed (Participants) | 17 | 15
Lesions
  Inflammatory Lesions | 4.03 (3.59) | 5.13 (5.77)
  Non-inflammatory Lesions | 7.29 (5.30) | 7.73 (8.17)

3. Secondary Outcome: Subject Improvement Assessment in Treatment Area Appearance
Description: Improvement as evaluated by subject using the Global Aesthetic Improvement Scale (GAIS) at 6 weeks after last treatment as compared to baseline where 3 = Very Much Improved, 2 = Much Improved, 1 = Improved, 0 = No Change, -1 = Worse, -2 = Much Worse and -3 = Very Much Worse.
Time Frame: Week 10 (6 weeks after last treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Diamondpolar Applicator, AC Dual Applicator | AC Dual Applicator
Number analyzed (Participants) | 18 | 17
Participants
  Much Worse (-2) | 1 | 0
  No Change (0) | 3 | 2
  Improved (1) | 10 | 9
  Much Improved (2) | 4 | 6

4. Secondary Outcome: Subject Assessment of Pain and Discomfort Associated With Treatments
Description: Pain and discomfort evaluated by subject using the 10 cm Visual Analog Scale where 0 cm is 'no pain' and 10 cm is 'intolerable pain'.
Time Frame: Immediately after each applicator treatment at Week 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diamondpolar Applicator, AC Dual Applicator | AC Dual Applicator
Number analyzed (Participants) | 18 | 19
units on a scale | 1.85 (1.68) | 2.53 (1.41)

5. Secondary Outcome: Subject Satisfaction With Treatment Outcome
Description: Satisfaction evaluated by subject using a 5-point Likert Scale where 4 = Very Satisfied, 3 = Satisfied, 2 Having No Opinion, 1 = Unsatisfied and 0 = Very Unsatisfied.
Time Frame: Week 10 (6 weeks after last treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Diamondpolar Applicator, AC Dual Applicator | AC Dual Applicator
Number analyzed (Participants) | 18 | 17
Participants
  Very Unsatisfied (0) | 0 | 1
  Unsatisfied (1) | 2 | 0
  Having No Opinion (2) | 2 | 4
  Satisfied (3) | 9 | 7
  Very Satisfied (4) | 5 | 5

6. Secondary Outcome: Subject Assessment of Improvement in Acne Related 'Quality of Life'
Description: Subject evaluated quality of life measured with the Acne Related Quality of Life Questionnaire at baseline where the total score varies from 0 to 114 with higher scores reflecting better quality of life.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diamondpolar Applicator, AC Dual Applicator | AC Dual Applicator
Number analyzed (Participants) | 20 | 19
score on a scale | 90.9 (29.12) | 85.47 (31.92)

7. Secondary Outcome: Subject Assessment of Pain and Discomfort Associated With Treatments
Description: as for outcome 4
Time Frame: Immediately after each applicator treatment at Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diamondpolar Applicator, AC Dual Applicator | AC Dual Applicator
Number analyzed (Participants) | 16 | 16
units on a scale | 2.30 (2.17) | 2.45 (1.60)

8. Secondary Outcome: Subject Assessment of Improvement in 'Quality of Life'
Description: Subject evaluated quality of life measured with the Acne Related Quality of Life Questionnaire at week 10 where the total score varies from 0 to 114 with higher scores reflecting better quality of life.
Time Frame: Week 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diamondpolar Applicator, AC Dual Applicator | AC Dual Applicator
Number analyzed (Participants) | 17 | 15
score on a scale | 113.29 (24.36) | 107.27 (32.84)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from time after informed consent was obtained until 7 days (for non-serious adverse events) and 30 days for serious adverse events after the last day of study participation, approximately 11 weeks for non-serious adverse events and 14 weeks for serious adverse events.
Arm/Group | Diamondpolar Applicator, AC Dual Applicator | AC Dual Applicator
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 2/20 | 2/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diamondpolar Applicator, AC Dual Applicator (N=20) | AC Dual Applicator (N=19)
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Subject did not complete the study as developed skin hypopigmentation post treatment.
Thermal burn (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-04): https://cdn.clinicaltrials.gov/large-docs/28/NCT02924428/Prot_SAP_000.pdf